CLINICAL TRIAL: NCT01298518
Title: A Phase 1B, Randomized, Double-Blind, Placebo-Controlled Trial To Assess The Efficacy And Safety Of 4-Week Administration Of Multiple Oral Doses Of PF-04620110 In Type 2 Diabetes Mellitus Subjects With Insufficient Glycemic Control On Metformin
Brief Title: A Multiple Dose Study Of PF-04620110 In Type 2 Diabetes Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B0961007
Record Dates: First submitted 2011-01-28; First posted 2011-02-17 (Estimated); Results first posted 2012-11-06 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes Patients
Keywords: multiple dose study in type 2 diabetes patients
MeSH Terms: interventions — PF-04620110

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04620110 (Experimental)
  Interventions: Drug: PF-04620110
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04620110 — 5 mg of PF-04620110 given once daily
  Arms: PF-04620110
Drug: PF-04620110 — 2.5 mg of PF-04620110 given twice daily
  Arms: PF-04620110
Drug: Placebo — Matching placebo giving for 4 weeks
  Arms: placebo

SUMMARY:
PF-04620110 is a novel compound proposed for the treatment of Type 2 diabetes mellitus. The primary purpose of this trial is to evaluate the safety and tolerability, and pharmacodynamics, of multiple oral doses of PF-04620110 in T2DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects between the ages of 18 and 60 years;
* Body Mass Index (BMI) of >25.0 kg/m2 and <40 kg/m2;
* Subjects must have a historical diagnosis of T2DM in accordance with the ADA guidelines;
* Subjects who have been on well-tolerated and stable doses of metformin

Exclusion Criteria:

* Recent evidence (6 months prior to screening) or history of unstable major organ disease;
* Diagnosis of Type 1 diabetes mellitus;
* Current medical history of myocardial infarction, unstable angina, or history of stroke (including TIA) within 6 months prior to Screening;
* Treatment with thiazolidinediones (TZDs), or subcutaneously administered antidiabetic agents;

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Chula Vista, California
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Miami Gardens, Florida

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961007&StudyName=A%20Multiple%20Dose%20Study%20Of%20PF-04620110%20In%20Type%202%20Diabetes%20Patients

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID: PF-04620110 2.5 milligram (mg) orally once daily (QD) in the morning and matching placebo orally once daily (QD) in the evening for Week 1 and 2, followed by PF-04620110 2.5 mg orally twice daily (BID) for Week 3 and 4.
- PF-04620110 5 mg QD: PF-04620110 5 mg orally once daily (QD) in the morning and matching placebo orally once daily (QD) in the evening for 4 weeks.
- Placebo: Matching placebo orally twice daily (BID) for 4 weeks.
Period: Overall Study
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Started | 16 | 16 | 16
Completed | 16 | 16 | 15
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 51.1 (5.8) | 53.4 (4.2) | 52.6 (6.3) | 52.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 4 | 13
  Male | 11 | 12 | 12 | 35
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (3.8) | 30.3 (3.3) | 32.6 (3.7) | 31.6 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Post-Prandial Glucose Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) After a Mixed Meal Tolerance Test (MMTT) at Day 28
Description: Change from baseline in post-prandial area under the plasma glucose concentration time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 post-MMTT glucose area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg*hr/dL
  Baseline (n=16, 16, 16) | 1052.7 (258.2) | 954.7 (249.2) | 1005.4 (190.0)
  Change at Day 28 (n=15, 16, 15) | -118.3 (269.0) | -143.0 (235.8) | -117.7 (157.4)

2. Secondary Outcome: Change From Baseline in 24-Hour Average Plasma Glucose (APG) Post-Dose at Day 28
Description: APG= AUC (0-24)/24. AUC (0-24) was computed using Linear trapezoidal method.
Time Frame: Baseline (Day -1); 24 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 APG value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg/dL
  Baseline (n=16, 16, 16) | 204.9 (52.2) | 188.0 (53.2) | 187.2 (36.5)
  Change at Day 28 (n=15, 16, 15) | -25.4 (60.9) | -23.4 (42.5) | -18.3 (29.6)

3. Secondary Outcome: Change From Baseline in Post-Prandial Insulin Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) After a Mixed Meal Tolerance Test (MMTT) at Day 28
Description: Change from baseline in post-prandial plasma insulin AUC under the plasma insulin concentration versus time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 post-MMTT insulin area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: micro-IU*hr/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
micro-IU*hr/mL
  Baseline (n=16, 16, 16) | 122.9 (82.9) | 220.2 (282.9) | 156.7 (63.3)
  Change at Day 28 (n=15, 16, 15) | 12.4 (63.9) | 0.6 (159.3) | 41.0 (46.0)

4. Secondary Outcome: Change From Baseline in Post-Prandial C-Peptide Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) After a Mixed Meal Tolerance Test (MMTT) at Day 28
Description: Change from baseline in post-prandial area under the plasma C-peptide concentration time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 post-MMTT C-peptide area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
ng*hr/mL
  Baseline (n=16, 16, 16) | 17.8 (6.2) | 21.6 (10.1) | 20.3 (5.4)
  Change at Day 28 (15, 16, 15) | -0.2 (6.0) | -4.0 (6.2) | -0.2 (5.2)

5. Secondary Outcome: Change From Baseline in Post-Prandial Net Triglyceride Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) After a Mixed Meal Tolerance Test (MMTT) at Day 28
Description: Change from baseline in post-prandial area under the plasma net triglyceride concentration time curve as determined by standardized MMTT. Linear trapezoidal method was used to compute AUC.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 post-MMTT net triglyceride area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg*hr/dL
  Baseline (n=16, 16, 16) | 860.6 (456.9) | 1014.4 (403.5) | 961.2 (380.7)
  Change at Day 28 (n=13, 16, 15) | -185.0 (436.7) | -100.5 (268.4) | -110.3 (245.3)

6. Secondary Outcome: Change From Baseline in Total Amide Glucagon Like Peptide-1 (GLP-1) and Active Glucagon Like Peptide-1 (GLP-1) Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) at Day 28
Description: Change from baseline in total amide GLP-1 and active GLP-1 area under the plasma concentration time curve was computed by Linear trapezoidal method.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 total amide GLP-1 and active GLP-1 area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: pmol*hr/L
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 15
pmol*hr/L
  Total amide GLP-1: Baseline (n=16, 15, 15) | 54.4 (26.8) | 63.2 (36.4) | 70.2 (88.1)
  Total amide GLP-1: Change at Day 28 (n=15, 15, 14) | 25.3 (27.9) | 4.7 (29.5) | -17.5 (88.9)
  Active GLP-1: Baseline (n=15, 16, 15) | 16.3 (11.5) | 21.0 (21.5) | 13.9 (11.4)
  Active GLP-1: Change at Day 28 (n=14, 14, 14) | 12.5 (15.0) | -0.5 (23.6) | 2.1 (11.1)

7. Secondary Outcome: Change From Baseline in Gastric Inhibitory Peptide (GIP) Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) at Day 28
Description: Change from baseline in GIP area under the plasma concentration time curve was computed by Linear trapezoidal method.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 GIP area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 15 | 16 | 16
pg*hr/mL
  Baseline (n=15, 16, 16) | 1372.8 (617.2) | 1181.0 (614.6) | 1619.2 (627.7)
  Change at Day 28 (n=14, 16, 15) | -141.6 (726.1) | -277.1 (541.4) | 46.8 (473.1)

8. Secondary Outcome: Change From Baseline in Peptide YY (PYY) Area Under the Concentration-Time Curve From Time 2 to 6 Hours (AUC 2-6) at Day 28
Description: Change from baseline in PYY area under the plasma concentration time curve was computed by Linear trapezoidal method.
Time Frame: Baseline (Day -1); 2 to 6 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 PYY area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 15 | 16 | 16
pg*hr/mL
  Baseline (n=15, 16, 16) | 409.0 (192.4) | 540.7 (273.8) | 395.0 (114.6)
  Change at Day 28 (n=14, 16, 14) | 196.6 (242.8) | 96.7 (194.2) | 24.4 (126.9)

9. Secondary Outcome: Change From Baseline in Fasting Glucose at Day 28
Time Frame: 0 hour (pre-dose) on Day -1, Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 fasting glucose value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg/dL
  Baseline (n=16, 16, 16) | 197.2 (54.6) | 180.9 (54.7) | 194.4 (37.4)
  Change at Day 28 (16, 16, 15) | -46.9 (49.5) | -27.1 (34.9) | -25.2 (32.1)

10. Secondary Outcome: Change From Baseline in Fasting Insulin at Day 28
Time Frame: 0 hour (pre-dose) on Day -1, Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 fasting insulin value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: micro-IU/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 9 | 10 | 8
micro-IU/mL
  Baseline (n=9, 10, 8) | 10.2 (6.9) | 19.8 (27.2) | 9.2 (4.2)
  Change at Day 28 (n=8, 9, 8) | -0.8 (4.0) | -8.0 (12.8) | 0.2 (2.7)

11. Secondary Outcome: Change From Baseline in Fasting Net Triglycerides at Day 28
Time Frame: 0 hour (pre-dose) on Day -1, Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 fasting net triglycerides value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg/dL
  Baseline (n=16, 16, 16) | 189.1 (111.7) | 234.8 (116.7) | 187.4 (81.6)
  Change at Day 28 (16, 16, 15) | -31.2 (103.6) | -18.4 (52.1) | -19.2 (56.7)

12. Secondary Outcome: Change From Baseline in Post-Lunch Glucose Excursions Area Under the Concentration-Time Curve From Time 6 to 10 Hours (AUC 6-10) Post-dose at Day 28
Description: Change from baseline in post-lunch glucose excursion under the plasma concentration time curve was computed by Linear trapezoidal method.
Time Frame: Baseline (Day -1); 6 to 10 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 post-lunch glucose excursion area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg*hr/dL
  Baseline (n=16, 16, 16) | 853.4 (293.4) | 772.3 (259.3) | 730.2 (174.9)
  Change at Day 28 (n=15, 16, 15) | -34.9 (377.2) | -41.4 (202.9) | -90.4 (157.3)

13. Secondary Outcome: Change From Baseline in Post-Dinner Glucose Excursions Area Under the Concentration-Time Curve From Time 12 to 16 Hours (AUC 12-16) Post-dose at Day 28
Description: Change from baseline in post-dinner glucose excursion under the plasma concentration time curve was computed by Linear trapezoidal method.
Time Frame: Baseline (Day -1); 12 to 16 hours post-dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 post-dinner glucose excursion area under the curve (AUC) value. Here, 'n' is participants evaluable at specified time points for each group.
Measure: Mean (Standard Deviation); unit: mg*hr/dL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Number analyzed (Participants) | 16 | 16 | 16
mg*hr/dL
  Baseline (n=16, 16, 16) | 851.2 (217.2) | 763.9 (215.8) | 759.4 (180.0)
  Change at Day 28 (n=15, 16, 15) | -132.8 (267.5) | -104.8 (210.8) | -41.4 (124.0)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-04620110
Time Frame: 24 hours post-morning dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 Cmax value.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD
Number analyzed (Participants) | 15 | 16
ng/mL | 91.0 (39.3) | 112.0 (43.7)

15. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) of PF-04620110
Time Frame: 24 hours post-morning dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 Cmin value.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD
Number analyzed (Participants) | 15 | 16
ng/mL | 16.2 (12.4) | 5.2 (9.2)

16. Secondary Outcome: Time to Cmax (Tmax) of PF-04620110
Time Frame: 24 hours post-morning dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 Tmax value.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD
Number analyzed (Participants) | 15 | 16
hr | 3.0 [1.7 to 12.0] | 3.0 [1.7 to 12.0]

17. Secondary Outcome: Area Under the Concentration-Time Curve AUC (0-24) of PF-04620110
Description: Area under the plasma concentration-time curve from time 0 (pre-dose) to 24 hours.
  AUC (0-24) was computed using the linear trapezoidal method.
Time Frame: 24 hours post-morning dose on Day 28
Population: Analysis population included all enrolled participants who received at least 1 dose of study medication and had at least 1 AUC(0-24) value.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD
Number analyzed (Participants) | 15 | 16
ng*hr/mL | 1055 (397.7) | 1027 (441.6)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID | PF-04620110 5 mg QD | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 12/16 | 15/16 | 10/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04620110 2.5 mg QD, Then PF-04620110 2.5 mg BID (N=16) | PF-04620110 5 mg QD (N=16) | Placebo (N=16)
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 3 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 7 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 6 | 0
Asthenia (General disorders) | 2 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 6 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.